CLINICAL TRIAL: NCT04472312
Title: Portal Pressure Effects of Phlebotomy Combined to Vasopressin Use in Cirrhotic Patients Undergoing Liver Transplantation: the PORTAL Study.
Brief Title: Portal Pressure Effects of Phlebotomy Combined to Vasopressin Use in Cirrhotic Patients Undergoing Liver Transplantation
Acronym: PORTAL
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 20.121
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Liver Transplantation; Portal Hypertension; Blood Transfusion; Blood Loss, Surgical
MeSH Terms: conditions — Hypertension, Portal; Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhotic patients undergoing a liver transplantation: The investigators aim to conduct a prospective observational, non-interventional study including all cirrhotic patients undergoing a liver transplantation with a planned use of vasopressin during the surgery.

SUMMARY:
Liver transplantation is the standard treatment for chronic advanced liver disease, whether or not associated with a primary liver tumor. The intraoperative bleeding and the need for blood transfusion, encountered in this major surgery are associated with increased morbidity and mortality. However, this hemorrhagic risk has been drastically reduced in the last 20 years and liver transplants without the use of blood products are now possible. Indeed, improvements in medical and surgical techniques associated with a better understanding of the pathophysiology of the cirrhotic patient have enabled this advance. One of the targeted therapeutic strategies is the control of portal hypertension. Several treatments have been sought, such as the use of splanchnic vasoconstrictors (such as vasopressin) and hypovolemic phlebotomy. These techniques reduce portal pressure and seem to reduce intraoperative bleeding with, even, a protective effect on kidney function. Their single-use or their combination is currently used in certain centers of expertise in liver transplantation. However, the hemodynamic effects of the combination of these 2 treatments on portal pressure has never been demonstrated. In this study, the effect of vasopressin, combined with a hypovolemic phlebotomy, on portal pressure in cirrhotic patients undergoing liver transplantation will be evaluated.

DETAILED DESCRIPTION:
METHODS

Objectives

The primary objective will be to measure the hemodynamic effects of vasopressin on portal pressure in cirrhotic patients who have had a hypovolemic phlebotomy during a liver transplant.

The secondary objectives will be to measure the effects of vasopressin on portal pressure in patients who have not had a phlebotomy and to compare this effect between patients who have or have not had a hypovolemic phlebotomy.

The tertiary objective will be to assess the effect of the variation in portal pressure under vasopressin, associated or not with a hypovolemic phlebotomy, on hemorrhagic clinical outcomes (intraoperative bleeding and blood transfusions).

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients undergoing a liver transplantation
* 18 years and older
* Planned use of vasopressin during the surgery

Exclusion Criteria:

* Fulminant or sub-fulminant hepatitis without underlying chronic liver disease
* Anesthetic plan does not include the use of vasopressin (contraindication or not relevant according to the anesthesiologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to conduct a prospective observational, non-interventional study, respecting current practice. This study will take place at the Centre de recherche de l'Université de Montréal (CHUM) where there are approximately 70 to 80 liver transplants per year.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Portal pressure measurement | During the surgery (intraoperatively)
  The venous pressure in the liver will be measured by inserting a very fine needle in the portal vein. The needle will be connected to a pressure sensor and will be removed after the measurement. This measure will be performed at three different moments during the surgery; 1) as soon as possible after the incision; 2) 5 minutes after the end of the hypovolemic phlebotomy (if performed); 3) 10 minutes after the start of vasopressin infusion.

SECONDARY OUTCOMES:
Intraoperative blood loss | At the end of the surgery
  During the liver transplantation, a cell salvage device (Cell Saver) will be set up in the operating room. As the surgery progresses, the blood lost by the patient will be collected using suctions. The volume of blood (mL) in the suctions will be measured at the end of the surgery, before the blood is cleaned and returned back to the patient.
Packed red blood cell transfusion rates | Intraoperatively and up to 24 hours following surgery
  Number of units of packed red blood cells transfused to participants will be recorded.
Rate of acute kidney injury (AKI) grade 2 or 3 | Assessed at 24 hours and 48 hours following surgery
  The onset or worsening of acute postoperative grade 2 or 3 renal failure according to KDIGO-AKI criteria.
Rate of new renal therapy replacement | Postoperative setting up to 7 days following surgery
  Any need of new renal therapy replacement occurring during the hospital stay up to 7 days following surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: François-Martin Carrier, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided